CLINICAL TRIAL: NCT02603588
Title: Effects of Sphenopalatine Ganglion Acupuncture on Nasal Ventilation and Autonomic Nervous Activity in Healthy Volunteers
Brief Title: The Effects of Sphenopalatine Ganglion Acupuncture on Nasal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Luo Zhang, Director, Beijing Institute of Otolaryngology., Beijing Tongren Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TR-acupuncture-1
Record Dates: First submitted 2015-11-07; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: Acupuncture; Sphenopalatine ganglion; Nasal ventilation; Neuropeptides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active acupuncture (Experimental): intervention: subjects in the active acupuncture group received active sphenopalatine ganglion acupuncture
  Interventions: Procedure: active sphenopalatine ganglion acupuncture
- sham acupuncture (Sham Comparator): intervention: subjects in the sham acupuncture group received sham sphenopalatine ganglion acupuncture
  Interventions: Procedure: sham sphenopalatine ganglion acupuncture

INTERVENTIONS:
Procedure: active sphenopalatine ganglion acupuncture — The acupuncture point was selected in the sphenopalatine ganglion (unilateral side). The acupuncture needle was inserted from the lower border of the zygomatic arch, slightly posterior to the suture protuberance between the zygomatic process and temporal process. The needle was rotated until the participant felt "de-qi" sensations.
  Arms: active acupuncture
Procedure: sham sphenopalatine ganglion acupuncture — The acupuncture point was selected same to the sphenopalatine ganglion. But the needle was inserted at the selected acupuncture site to a depth of only 2-3cm, and the procedure of rotating, twirling and thrusting the needle was repeated, in order to blind the subject to the sham treatment.
  Arms: sham acupuncture

SUMMARY:
Sphenopalatine ganglion (SPG)-acupuncture has been shown to exhibit distinct effects in treatment of nasal inflammatory disease, but the mechanisms remain largely unknown. Investigators aimed to assess the effects of SPG acupuncture for nasal ventilation function and autonomic nervous system in health volunteers. The randomized, double-blind, controlled clinical trial enrolled healthy volunteers.Healthy subjects were randomly assigned to either active SPG-acupuncture group or sham-acupuncture group. All subjects were assessed for self-reported nasal ventilation, nasal patency (nasal airway resistance (NAR) and nasal cavity volume (NVC)), exhaled nasal nitric oxide (nNO) before and after acupuncture. Meanwhile, in order to explore underlying mechanisms of SPG acupuncture, the changes in neuropeptides (substance P (SP), vasoactive intestinal peptide (VIP) and neuropeptide Y (NPY)) in nasal secretions were investigated at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking volunteers
* without history of nasal disease (allergic rhinitis, sinusitis, nasal polyps, nasal septum deviation and history of nose surgery) or lung disease (asthma, chronic obstructive pulmonary disease and fibrosis)
* free of upper and lower respiratory tract infections for at least 4 weeks before beginning the study.
* negative skin prick test for allergy

Exclusion Criteria:

* had received acupuncture within the last four weeks before the start of the study
* no history of diabetes mellitus, autonomic neuropathy, coronary heart disease or hypertension.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The change of subjective perception nasal ventilation | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  The subjective perception of nasal ventilation was self-assessed by participants according to three categories: unchanged, better, and worse. Number of participants reported unchanged or better was analysed.

SECONDARY OUTCOMES:
The change of exhaled nasal nitric oxide assessed by nitric oxide analyser | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  A nitric oxide analyser was used to measure exhaled nasal nitric oxide (nNO). Briefly, NO-free air was aspirated through the nasal cavity at a flow rate of 50 ml/s. The subject exhaled against the air-resistance, resulting in an intraoral pressure to close the velum and prevent mixture of oral and nasal gas. Nasal gas from this circuit was continuously routed in part directly into the analyser for determination of nNO, and the level of nNO(ppb) was calculated from a plateau lasting for at least 3s.
The change of nasal patency assessed by acoustic rhinometry | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  Acoustic rhinometry was performed to measure the total nasal cavity volume (cm³).
The change of substance P in nasal secretions were analysed by Enzyme linked immunosorbent assay | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  Nasal secretions were obtained by inserting a postoperative sinus pack in the nasal cavity (acupuncture side) for five minutes. The quantity of secretions was determined by comparing the weight of the sponges before and after insertion and 2 ml of 0.9% sodium chloride solution was added to each sponge. The sponges were stored at 4°C for two hours and the nasal secretions were recovered from the sponges by centrifugation at 1500 g for 15 minutes at 4°C. The supernatants were separated and stored in aliquots at -20°C until further analysis. The levels of substance P(pg/ml) were analysed.
The change of nasal patency assessed by Rhinomanometer | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  Rhinomanometer was used to measure unilateral nasal airway resistance (Pa·cm-³·s-1) and the total nasal airway resistance.
The change of vasoactive intestinal peptide in nasal secretions were analysed by Enzyme linked immunosorbent assay | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  Nasal secretions were obtained by inserting a postoperative sinus pack in the nasal cavity (acupuncture side) for five minutes. The quantity of secretions was determined by comparing the weight of the sponges before and after insertion and 2 ml of 0.9% sodium chloride solution was added to each sponge. The sponges were stored at 4°C for two hours and the nasal secretions were recovered from the sponges by centrifugation at 1500 g for 15 minutes at 4°C. The supernatants were separated and stored in aliquots at -20°C until further analysis. The levels of vasoactive intestinal peptide (ng/ml) were analysed.
The change of neuropeptide Y in nasal secretions were analysed by Enzyme linked immunosorbent assay | at baseline, 30 minutes, 2 hours, and 24 hours after acupuncture
  Nasal secretions were obtained by inserting a postoperative sinus pack in the nasal cavity (acupuncture side) for five minutes. The quantity of secretions was determined by comparing the weight of the sponges before and after insertion and 2 ml of 0.9% sodium chloride solution was added to each sponge. The sponges were stored at 4°C for two hours and the nasal secretions were recovered from the sponges by centrifugation at 1500 g for 15 minutes at 4°C. The supernatants were separated and stored in aliquots at -20°C until further analysis. The levels of neuropeptide Y (pg/ml) were analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Institute of Otolaryngology
Locations (1):
- Beijing Tongren Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Shakeel M, Trinidade A, Ah-See KW. Complementary and alternative medicine use by otolaryngology patients: a paradigm for practitioners in all surgical specialties. Eur Arch Otorhinolaryngol. 2010 Jun;267(6):961-71. doi: 10.1007/s00405-009-1098-1. Epub 2009 Sep 22. PMID 19771443
- [Background] Pletcher SD, Goldberg AN, Lee J, Acquah J. Use of acupuncture in the treatment of sinus and nasal symptoms: results of a practitioner survey. Am J Rhinol. 2006 Mar-Apr;20(2):235-7. PMID 16686397
- [Background] Sertel S, Bergmann Z, Ratzlaff K, Baumann I, Greten HJ, Plinkert PK. Acupuncture for nasal congestion: a prospective, randomized, double-blind, placebo-controlled clinical pilot study. Am J Rhinol Allergy. 2009 Nov-Dec;23(6):e23-8. doi: 10.2500/ajra.2009.23.3380. Epub 2009 Sep 18. PMID 19769799
- [Background] Zhang L, Yang W, Wang KJ. [Acupuncture at ganglion pterygoplatinum for 71 cases of chronic simple rhinitis]. Zhongguo Zhen Jiu. 2013 Jun;33(6):495-6. No abstract available. Chinese. PMID 23967633
- [Background] Baraniuk JN, Merck SJ. Neuroregulation of human nasal mucosa. Ann N Y Acad Sci. 2009 Jul;1170:604-9. doi: 10.1111/j.1749-6632.2009.04481.x. PMID 19686200
- [Background] Loehrl TA. Autonomic dysfunction, allergy and the upper airway. Curr Opin Otolaryngol Head Neck Surg. 2007 Aug;15(4):264-7. doi: 10.1097/MOO.0b013e32826fbcc9. PMID 17620901
- [Background] McDonald JL, Cripps AW, Smith PK, Smith CA, Xue CC, Golianu B. The anti-inflammatory effects of acupuncture and their relevance to allergic rhinitis: a narrative review and proposed model. Evid Based Complement Alternat Med. 2013;2013:591796. doi: 10.1155/2013/591796. Epub 2013 Feb 14. PMID 23476696